CLINICAL TRIAL: NCT03309254
Title: Role of Glycaemic Index and High Protein Meal in Response of Blood Biomarkers for Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: University of Auckland, New Zealand (Other); Massey University (Other); Riddet University (Unknown)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015/01077
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Glycemic Index (Experimental): White Bread with Turkey breast meat (2 slices) Turkey Breast (7 slices) Chamomile Tea with 25 grams glucose Almonds 15 grams
  Interventions: Other: High Glycemic Index
- Low Glycemic Index (Experimental): Multi-grain Bread with Turkey breast meat (2 slices) Turkey Breast (6 slices) Chamomile Tea with 25 grams fructose Cashews 10 grams
  Interventions: Other: Low Glycemic Index

INTERVENTIONS:
Other: High Glycemic Index — High Glycemic Index Food
  Arms: High Glycemic Index
Other: Low Glycemic Index — Low Glycemic Index Food
  Arms: Low Glycemic Index

SUMMARY:
This study aims to demonstrate the effectiveness of increased protein ingestion, particularly when coupled with a low glycaemic index (GI) to reduce biomarkers related to high risk of diabetes.

DETAILED DESCRIPTION:
A randomized cross-over study and subjects will be randomized to take either the high GI or low GI meal. The sequence of the meal will be generated using an online randomiser generator.During screening administer informed consent.Measure height, weight, waist and hip circumference.Blood draw: Two fingerpricks, 5 minutes apart. 1 X 10ml red tube top to prepare serum. Serum and red platelets into separate microtubes. Serum will be used to analyse fasting blood glucose, lipid profile, C-Reactive Protein (CPR), insulin and apolipoprotein. Red platelets will be stored separately for DNA genotyping. During the study visits,On Day 1, subjects will come to the Centre at around 4:00 pm to have the continuous glucose monitoring (CGMS) system inserted. CGMS will be used to measure 24 hour blood glucose concentrations. The sensor records interstitial blood glucose concentrations every five minutes. This will involve the insertion of a small sensor under the skin in the abdomen, which will be carried out by using a device that produces minimal pain and discomfort.Subjects will have to wait in the laboratory for one hour after insertion for the sensor to be stabilized. After one hour the inserted CGMS sensor will be calibrated against a manual finger-prick blood glucose sample.Manual calibration using finger-prick blood samples will need to be carried out before every meal and before bed in the night. The calibrations before dinner and bed will have to be carried out by the subjects at home.Therefore, the subjects will be provided with a finger-prick blood glucose test kit to take home and instructed on how to correctly use it and measure blood glucose values. Subjects will then consume the standardised dinner at around 7pm.Subjects will be asked to fast overnight and instructed to avoid eating or drinking anything, except water, after 10pm. Subjects will arrived between 8.00am and 8.30am the following morning. Baseline blood samples will be collected. A venous cannula will be inserted and a fasting blood sample collected. Baseline basal metabolic rate will be measured using hood-ventilated indirect calorimetry for 30mins during fasting. Subjects will then consume the test meal. Further venous blood samples will be collected at regular intervals for up to 4hours postprandial. After meal, subjects will enter the hood-ventilated indirect calorimetry and measure post-prandial respiratory quotient for 4 hours. A medium GI lunch will then be provided and the subject can either stay in the centre or return to the centre 4 hours after lunch to remove the CGMS.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 55-70 years old, 5 years post-menopausal (a: healthy, b: fasting blood glucose, ≥5.1mmol/l) or
* Group 2: 23-54 years old (a: healthy, b: fasting blood glucose, ≥5.1mmol/l)
* Body mass index between 18 and 30 kg/m2

Exclusion Criteria:

* Have family history of diabetes or any major chronic disease such as diabetes, heart disease or cancer
* On prescribed medication known to affect blood glucose concentrations or major effects on body fat distribution
* Have allergic/intolerant to any of the test foods (e.g bread, turkey breast, almond, cashew, glucose, fructose and chamomile tea.
* Have gastrointestinal diseases that may interfere with digestion or nutrient absorption
* Have medical or surgical events requiring hospitalization within the preceding three months
* Currently pregnant or breastfeeding
* Have G6PD deficiency

Ages: 23 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All female subjects
Enrollment: 46 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Glycemic response | up to 8 hours
  measured using continuous glucose monitoring system
Glycemic response | up to 4 hours
  measured using COBAS Analyzer

SECONDARY OUTCOMES:
Blood Biochemistry | up to 4 hours
  measured using COBAS Analyzer
Respiratory quotient and fat oxidation | up to 4 hours
  measured using indirect calorimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camps SG, Koh HR, Wang NX, Henry CJ. High fructose consumption with a high-protein meal is associated with decreased glycemia and increased thermogenesis but reduced fat oxidation: A randomized controlled trial. Nutrition. 2019 Feb;58:77-82. doi: 10.1016/j.nut.2018.06.024. Epub 2018 Jul 20. PMID 30391694